CLINICAL TRIAL: NCT07109687
Title: Comparison of the Effects of High-Intensity Interval Training and Moderate-Intensity Continuous Training on Peripheral and Respiratory Muscle Oxygenation, Pulmonary Function, Exercise Capacity, and Peripheral Muscle Strength in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: HIIT Versus MICT in COPD: Effects on Oxygenation, Pulmonary Function, and Strength
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aynur Demirel (Other)
Collaborators: Antalya Bilim University (Other); Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSV-000021
Record Dates: First submitted 2025-07-16; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: High Intensity Interval Training; Exercise Training; Muscle Oxygenation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: HIIT or MICT will be applied in patients with COPD groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Statistical Analyzer will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): standard aerobic exercise will apply in moderate intensity continuous training.
  Interventions: Other: MICT
- interval exercise group (Experimental)
  Interventions: Other: HIIT GROUP

INTERVENTIONS:
Other: HIIT GROUP — Participants will perform a 31-minute protocol on a cycle ergometer consisting of 1-minute high-intensity intervals at 90% of peak workload (W peak) and low-intensity intervals at 30-40% of W peak, twice a week for 8 weeks.
  Arms: interval exercise group
Other: MICT — Moderate intensity continous exercise
  Arms: Control Group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive condition marked by airflow limitation and chronic inflammation, leading to reduced exercise capacity, peripheral muscle dysfunction, and dyspnea. High-Intensity Interval Training (HIIT) may offer a promising alternative for patients with low exercise tolerance; however, evidence on its effectiveness remains limited.

This study aims to compare the effects of HIIT and Moderate-Intensity Continuous Training (MICT) on muscle oxygenation, pulmonary function, exercise capacity, and peripheral muscle strength in individuals with COPD. Participants will undergo an 8-week exercise program, twice weekly. HIIT will consist of 1-minute intervals at 90% and 30-40% of peak workload, while MICT will involve continuous cycling at 65% of peak workload. Outcomes will be assessed at baseline, week 4, and week 8. Data will be analyzed using SPSS. This study seeks to determine the more effective training modality to optimize COPD rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Chronic Obstructive Pulmonary Disease (COPD),
* GOLD stage 2, 3, or 4,
* Willing to participate in the study,
* Aged between 40 and 80 years,
* Clinically stable (no significant deterioration in the current medical condition, no recent initiation of a new treatment, and no complications requiring hospitalization).

Exclusion Criteria:

* Presence of visual, auditory, vestibular, cognitive, or neurological impairments that may affect balance,
* Any orthopedic, neurological, or cardiac conditions that may interfere with study participation or exercise,
* Presence of serious chronic diseases such as congestive heart failure, coronary artery disease, or chronic renal failure,
* Conditions that may cause physical limitations (e.g., limb amputation, significant musculoskeletal disorders, or postural abnormalities such as kyphosis or lordosis).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral and Respiratory Muscle Oxygenation | at the baseline, at the 4th week, at the end of the 8th week.
  Muscle oxygenation will be measured using Near-Infrared Spectroscopy from the dominant quadriceps (peripheral) and 7th intercostal space (respiratory) during rest, warm-up, exercise, recovery phases, and 5 minutes post-exercise. Parameters include SmO₂_basal, SmO₂_max, SmO₂_min, SmO₂_maxrec, ∆SmO₂_max, SmO₂_deox, SmO₂_reoxy, and ∆SmO₂_maxrec.

SECONDARY OUTCOMES:
Pulmonary Function test | at the baseline, at the 4th week, at the end of the 8th week.
  Pulmonary function will be evaluated using spirometry in accordance with ATS/ERS guidelines. the outcomes presented as liter/minute.
Functional Exercise Capacity | at the baseline, at the 4th week, at the end of the 8th week.
  Functional exercise capacity will be assessed using the 6-Minute Walk Test (6MWT) according to ATS guidelines.
Dyspnea | at the baseline, at the 4th week, at the end of the 8th week.
  Dyspnea will be assessed using the Modified Medical Research Council (mMRC) Dyspnea Scale, a 5-point ordinal scale evaluating activity-induced breathlessness.
Upper extremity Muscle Strength | at the baseline, at the 4th week, at the end of the 8th week.
  Upper extremity will measure by hand dynomometer. The highest grip force will be recorded as kilograms.
Activities of Daily Living | at the baseline, at the 4th week, at the end of the 8th week.
  Activity limitation due to dyspnea will be assessed by the London Chest Activity of Daily Living Scale (LCADL). Total and subscale scores will be analyzed (range: 0-75).
Health-Related Quality of Life | at the baseline, at the 4th week, at the end of the 8th week.
  Quality of life will be evaluated using the St. George's Respiratory Questionnaire (SGRQ). Total and subscale scores (Symptoms, Activity, Impacts) will be recorded (range: 0-100).
Comorbidities | at the baseline, at the 4th week, at the end of the 8th week.
  Comorbidity burden will be assessed using the Charlson Comorbidity Index (CCI)
lower extremity endurance test | at baseline, at the 4th week and at the end of 8th week.
  30 second chair stand test will use. The number of repetitions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Fulsen Bozkus, MD., Prof., Study Director — Sağlık Bilimleri University Antalya Health Application and Research Center; Aynur Demirel, PT, PhD, Assoc. Prof., Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided